CLINICAL TRIAL: NCT00392080
Title: A Multicenter, Randomized, Placebo And Active-Controlled Study Of The Effect Of CJ-023,423 On The Incidence Gastroduodenal Endoscopic Ulcers In Healthy Subjects
Brief Title: A Study Of The Effect Of CJ-023,423 On The Incidence Of Stomach Ulcers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5231018
Record Dates: First submitted 2006-10-23; First posted 2006-10-25 (Estimated); Last update posted 2008-03-24 (Estimated); Status verified 2008-03

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — grapiprant; Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 3 (Placebo Comparator)
  Interventions: Drug: placebo
- 1 (Experimental): 75 mg BID
  Interventions: Drug: naproxen
- 2 (Experimental)
  Interventions: Drug: CJ-023,423

INTERVENTIONS:
Drug: CJ-023,423 — 75 mg BID
  Arms: 2
Drug: placebo — placebo
  Arms: 3
Drug: naproxen — naproxen
  Arms: 1

SUMMARY:
CJ-023,423 is a new medication being developed as an anti-inflammatory agent for the treatment of the signs and symptoms of osteoarthritis (OA). The purpose of this study is to evaluate whether patients treated with CJ-023,423 for 7 days (14 doses) have fewer gastrointestinal ulcers compared to patients treated with naproxen and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Is a healthy adult 18 to 75 years of age, inclusive; healthy is defined as no clinically relevant abnormalities identified as detailed medical history, full physical examination, including blood pressure [BP] and pulse rate [PR]measurement, 12-lead electrocardiogram [ECG], and clinical safety laboratory tests
* If female and of childbearing potential (includes women who have been postmenopausal for < 2 years ), must be using adequate contraception, must not be lactating and must have had a negative serum pregnancy test at Screening and a negative urine pregnancy test result within 24 hours prior to receiving study drug. The site investigator must ensure that female subjects are not pregnant prior to receiving the first dose of drug;

Exclusion Criteria:

* Endoscopic evidence of inflammation, ulceration, erosion, petechiae, or active bleeding in the esophagus, stomach, pyloric channel, or duodenum at the baseline/ randomization (Day 1) endoscopy (Mucosal Grading Scale score >0);
* Active GI disease (e.g. inflammatory bowel disease), a history of gastroduodenal ulcers or bleeding, or a history of any gastric or duodenal surgery;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2006-11; Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the presence of gastroduodenal ulcers in each subject, as determined by a UGI endoscopy at the end of the treatment | 7 days

SECONDARY OUTCOMES:
Incidence of treatment-emergent, all-causality GI body system adverse events | Duration of trial
Severity of Dyspepsia Assessment (SODA) | Duration of trial
Post treatment gastric, duodenal and gastroduodenal endoscopic scores (according to the mucosal grading scale). The gastroduodenal score is defined as the higher of the gastric and duodenal scores. | Duration of trial
Incidence of any gastric ulcer | Duration of trial
Incidence of any duodenal ulcer | Duration of trial
Incidence of any gastroduodenal erosion or ulcer | Duration of trial
Incidence of any gastric erosion or ulcer | Duration of trial
Incidence of any duodenal erosion or ulcer | Duration of trial
Incidence of any esophageal ulcer using the traditional grading method of: normal, erosion or ulcer | Duration of trial
Incidence of any esophageal ulcer or erosion using the LA classification: esophageal ulcers and erosions method with a Grade A, B, C, or D) | Duration of trial
Number of gastroduodenal ulcers in each subject | Duration of trial

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- United States (9):
  - Pfizer Investigational Site, Anaheim, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Jupiter, Florida
  - Pfizer Investigational Site, Ocoee, Florida
  - Pfizer Investigational Site, South Miami, Florida
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Chesapeake, Virginia

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5231018&StudyName=A%20Study%20Of%20The%20Effect%20Of%20CJ-023%2C423%20On%20The%20Incidence%20Of%20Stomach%20Ulcers